CLINICAL TRIAL: NCT02807077
Title: A Phase 1 Open-Label, Single-Dose, Parallel-Group Study to Determine the Pharmacokinetics of Pacritinib in Patients With Mild, Moderate, and Severe Renal Impairment and End-Stage Renal Disease (ESRD) Compared to Healthy Subjects
Brief Title: PK of Pacritinib in Patients With Mild, Moderate, Severe Renal Impairment and ESRD Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAC105
Record Dates: First submitted 2016-05-03; First posted 2016-06-21 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Myelofibrosis
Keywords: Healthy subjects
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

ARMS (5):
- Subjects with mild renal impairment (Experimental): Group 1, will consist of patients each with mild, moderate, or severe renal disease, respectively, based on their estimated glomerular filtration rate (eGFR, calculated by the Modification of Diet in Renal Disease [MDRD] study equation). Each of these patients will receive a single 400 mg dose of pacritinib.
  Interventions: Drug: Pacritinib
- Subjects with moderate renal impairment (Experimental): Group 2, will consist of patients each with mild, moderate, or severe renal disease, respectively, based on their estimated glomerular filtration rate (eGFR, calculated by the Modification of Diet in Renal Disease [MDRD] study equation). Each of these patients will receive a single 400 mg dose of pacritinib.
  Interventions: Drug: Pacritinib
- Subjects with severe renal impairment (Experimental): Group 3, will consist of patients each with mild, moderate, or severe renal disease, respectively, based on their estimated glomerular filtration rate (eGFR, calculated by the Modification of Diet in Renal Disease [MDRD] study equation). Each of these patients will receive a single 400 mg dose of pacritinib.
  Interventions: Drug: Pacritinib
- Subjects with ESRD (Experimental): Group 4, will consist of patients with ESRD requiring hemodialysis who have been on a stable dialysis regimen for at least 6 months. In this cohort only, patients will participate in 2 treatment periods, Dialysis and Inter-Dialysis, separated by a 14-day period between pacritinib administration. In the Dialysis Treatment Period, a single 400 mg dose of pacritinib will be administered 4 hours prior to each patient's normally scheduled hemodialysis. In the Inter-Dialysis Treatment Period, a single 400 mg dose of pacritinib will be administered immediately after the end of the patient's normally scheduled hemodialysis session.
  Interventions: Drug: Pacritinib
- Healthy subjects (Experimental): Group 5, will consist of 8 healthy subjects enrolled to match the sex-, age-, and weight of the patients with mild, moderate, and severe renal impairment and patients with ESRD enrolled in the study. Healthy subjects will be administered a single 400 mg dose of pacritinib.
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Group 1, 2, 3, and 5 will be administered single oral 400-mg dose of pacritinib. Subjects in the Group 4 received a single 400-mg dose of pacritinib during two different treatment periods: Dialysis and Inter-Dialysis

SUMMARY:
This is a Phase 1 open label, single dose, 5 parallel-group study in which a single 400 mg dose of pacritinib will be administered orally to patients with renal impairment (mild, moderate, severe, and patients with ESRD requiring hemodialysis) and sex-, age- and weight-matched healthy subjects.Patients with ESRD will receive a single 400 mg dose of pacritinib during 2 different treatment periods: Dialysis and Inter-Dialysis. The primary objective of the study is to evaluate the pharmacokinetics and safety of pacritinib in renal impairment.

DETAILED DESCRIPTION:
Groups 1, 2, and 3 will consist of 8 patients each with mild, moderate, or severe renal disease, respectively, based on their estimated glomerular filtration rate (eGFR, calculated by the Modification of Diet in Renal Disease [MDRD] study equation). Each of these patients will receive a single 400 mg dose of pacritinib.

Group 4 will consist of 8 patients with ESRD requiring hemodialysis who have been on a stable dialysis regimen for at least 6 months. In this cohort only, patients will participate in 2 treatment periods, Dialysis and Inter-Dialysis, separated by a 14-day period between pacritinib administration. In the Dialysis Treatment Period, a single 400 mg dose of pacritinib will be administered 4 hours prior to each patient's normally scheduled hemodialysis. In the Inter-Dialysis Treatment Period, a single 400 mg dose of pacritinib will be administered immediately after the end of the patient's normally scheduled hemodialysis session.

Group 5 will consist of 8 healthy subjects enrolled to match the sex-, age-, and weight of the patients with mild, moderate, and severe renal impairment and patients with ESRD enrolled in the study. Healthy subjects will be administered a single 400 mg dose of pacritinib.

ELIGIBILITY:
Inclusion Criteria:

All Study Participants

1. Male and/or female participants aged 18 to 85 years (inclusive)
2. Male, non-fertile female or female of childbearing potential using a medically approved birth control method

   * Females must be non-pregnant and non-lactating, and females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days, or agree to use contraception from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 30 days after Study Completion. One of the following forms of contraception must be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 14 days after the final dose administration: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (e.g.,NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1)
   * Males will be sterile, or completely abstain from sexual intercourse, or agree to use, from Check-in (Day -1) until 90 days following Study Completion/ET, one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; a contraceptive sponge with spermicide; an intravaginal system; a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives. Participants will refrain from sperm donation from Check-in (Day -1) until 90 days following Study Completion
3. Body mass index (BMI) 18-33kg/m2 (inclusive) at Screening
4. Negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in (Day - 1) for Groups 1-3 and 5. Negative test for selected drugs of abuse (including alcohol) is only required at Screening in Group 4
5. Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti HCV]) and negative human immunodeficiency virus (HIV) antibody screens
6. Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent. Legal authorized representatives are not permitted

   Patients with Renal Impairment Only

   In addition to the inclusion criteria specified for "All Study Participants" above, patients with renal impairment must meet the following criteria:
7. Have stable renal disease without evidence of progressive renal disease (i.e. no known significant change of eGFR for 12 weeks)

   * mild renal impairment: eGFR 60-89 mL/min/1.73 m2
   * moderate renal impairment: eGFR 30-59 mL/min/1.73 m2
   * severe renal impairment: CrCl from eGFR 15-29 mL/min/1.73 m2
   * ESRD: requiring dialysis and have been on a stable dialysis regimen for at least 6 months

   Renal function will be determined from Screening serum creatinine value using the MDRD Study equation
8. Vital signs (after 5 minutes resting measured in the supine position) within the following ranges as guidance for the Investigator:

   * oral body temperature between 35.0-37.8 °C
   * systolic blood pressure, 95-180 mm Hg
   * diastolic blood pressure, 55-95 mm Hg
   * pulse rate, 50-95 bpm

   Blood pressure and pulse will be taken again in a standing position. After 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mm Hg drop in diastolic blood pressure associated with symptomatic postural hypotension

   Healthy Subjects Only

   In addition to the inclusion criteria specified for "All Study Participants" above, healthy subjects must meet the following criteria:
9. No history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (e.g., celiac disease, peptic ulcer, gastro esophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator; appendectomy and cholecystectomy are not considered to be clinically significant disease)
10. Normal renal function, eGFR ≥90 mL/min/1.73m2 (determined by Screening serum creatinine using the MDRD Study equation)
11. Matched with all enrolled patients with renal impairment for age classes in the 0-25, 26-50, 51-75, and 76-100 percentiles of age distribution
12. Matched with all enrolled patients with renal impairment for weight (BMI) classes in the 0-25, 26-50, 51-75, and 76-100 percentiles of BMI distribution
13. Matched according to the sex distribution of all enrolled patients with renal impairment
14. Vital signs (after 5 minutes resting measured in the supine position) within the following ranges as guidance for the Investigator:

    * oral body temperature between 35.0-37.5 °C
    * systolic blood pressure, 90-160 mm Hg
    * diastolic blood pressure, 50-100 mm Hg
    * pulse rate, 45-90 bpm

Blood pressure and pulse will be taken again in a standing position. After 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mm Hg drop in diastolic blood pressure associated with symptomatic postural hypotension

Exclusion Criteria:

All Study Participants

Participants meeting any of the following criteria will be excluded from entry into or continuation in the study unless sponsor approval is obtained:

1. Pregnant or lactating female
2. Renal transplant at any time
3. Liver cirrhosis or a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result
4. History of immunodeficiency diseases, including a positive HIV antibody test result
5. Acute renal failure
6. History of chronic or recurrent urinary tract infection active within the past 30 days
7. History of pelvic irradiation within the past 30 days
8. Alcohol related hepatic disease
9. History of malignancy except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps
10. Any of the following within the past 6 months:

    * myocardial infarction (MI) (if the Screening ECG reveals patterns consistent with a MI and the date of the event cannot be determined, then the subject can enter the study at the discretion of the Investigator and/or local medical monitor, with sponsor's permission)
    * coronary artery bypass surgery or percutaneous coronary intervention
    * unstable angina or stroke
11. Past medical history of clinically significant ECG abnormalities, presence of an abnormal ECG (which in the Investigator's opinion is clinically significant), QTcF>450 msec, or has concomitant conditions that increase risk for QTc interval prolongation (e.g., heart failure, hypokalemia [defined as serum potassium <3.0mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome)
12. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
13. Any medical or surgical conditions that might significantly interfere with the gastrointestinal absorption, distribution, metabolism, or excretion of the investigational drug. This includes any history of a significant disease of the gastrointestinal tract, pancreas, liver, kidneys, and/or blood-forming organs. It does not include appendectomy, cholecystectomy, hernia repair, or underlying renal disease or abnormalities that occur as a direct result of renal disease in the renal impairment patients or abnormalities that occur as a direct result of renal disease
14. History of drug or alcohol abuse within the last 6 months, or evidence of recent drug or alcohol abuse as indicated by laboratory assays conducted during screening or baseline evaluations
15. Heavy use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) and during the entire study, defined as urinary cotinine > 150 ng/mL
16. Consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to screening and during the entire study
17. Consumption of grapefruit-containing foods and beverages or other potent cytochrome P450 (CYP)3A4 inhibitors or inducers for 7 days prior to Check-in (Day -1) and during the entire study
18. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1), whichever is longer, and during the entire study
19. Use of oral, implantable, injectable, or transdermal contraceptives within 10 days prior to Check-in (Day -1) or from the time of signing the informed consent (females only) until 14 days after the final dose administration
20. Use of any over-the-counter, non-prescription medications, vitamins, or minerals (except as prescribed by a physician), within 14 days prior to Check-in (Day -1) and during the entire study
21. Use of phytotherapeutic/herbal/plant-derived preparations within 14 days prior to Check-in (Day -1) of and during the entire study
22. Use of potent inducers of CYP3A4 within 30 days of Check-in (Day -1)
23. Use of potent inhibitors of CYP3A4 within 15 days of Check-in (Day -1)
24. Poor peripheral venous access
25. Donation or loss of 400 mL or more of blood or plasma within 8 weeks prior to Check-in (Day -1) and through entire study
26. Receipt of blood products within 2 months prior to Check-in (Day -1)
27. Any diarrhea or vomiting during the Screening period or at Check-in (Day -1)
28. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study
29. Any of the following concomitant medications within 30 days of Check-in (Day -1) (unless cited otherwise below):

    * potassium-sparing diuretics e.g. spironolactone, triamterene, amiloride (within 14 days of Check-in)
    * class Ia, Ib and Ic or III anti-arrhythmics
    * probenecid
    * any medication that is contraindicated in moderate or severe renally impaired population
    * any drug with a known and frequent toxicity to a major organ system within 3 months of Screening (i.e., cytostatic drugs)
30. Any of the following (repeated and confirmed) laboratory abnormalities at Screening or Check-in:

    * Clinically significant (as judged by the Investigator in consultation with the Sponsor) laboratory abnormalities except elevated blood urea nitrogen (BUN), elevated serum creatinine, hyperglycemia, and/or glycosuria
    * Alanine aminotransferase (ALT)>1.5xULN
    * Aspartate aminotransferase (AST)>1.5xULN
    * Total bilirubin >1.3x ULN (unless due to Gilbert's Syndrome)
    * Hemoglobin < 8 g/dL

    Laboratory testing may be repeated once prior to dosing (to rule out any possible laboratory error)
31. Planned surgery during the study period
32. Subjects who are deemed vulnerable by way of imprisonment, remand or detention

    Patients with Renal Impairment Only

    In addition to the exclusion criteria specified for "All Subjects" above, any patient with renal impairment who meets the following criteria will be excluded from entry into the study:
33. Any condition that would compromise patients' safety during study participation
34. Participants in Groups 1-3: Difficulty voiding or urinary tract obstruction at Check-in or undergoing any method of dialysis (hemodialysis, peritoneal dialysis)
35. Screening physical exam or ECG finding considered of clinical significance by the Investigator, or a laboratory evaluation outside of the normal reference range with the exception of values that are related to renal impairment
36. Any significant acute or chronic disease (except renal impairment) which is unstable or can interfere with the objectives of the study
37. Any change in stable dose regimens, either over-the-counter or prescription, for chronic medical conditions (e.g. diabetes, dyslipidemia, renal impairment) within 4 weeks preceding dosing

    Healthy Subjects Only

    In addition to the exclusion criteria specified for "All Study Participants" above, any healthy subject who meets the following criteria will be excluded from entry into the study:
38. Any screening or baseline physical exam, EKG, or laboratories outside the normal range and deemed clinically significant by the Investigator. Results deemed not clinically significant by the Investigator in consultation with the Sponsor are allowable.
39. Use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) and during the entire study
40. History of renal impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The time to reach maximum plasma concentration (tmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The apparent terminal elimination rate constant (λZ) and the respective apparent terminal elimination half-life (t½) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The apparent volume of distribution (Vd) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects
The apparent total body clearance (CL/F) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose. Urine- 0-168 hr interval
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule in patients with renal impairment and matched healthy subjects

SECONDARY OUTCOMES:
Incidence of Treatment emergent Adverse Events | Day 1 to Day 8
  Adverse events, vital signs, physical examinations, clinical laboratory evaluations, and ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Igor Codreanu, MD, Principal Investigator — Republican Clinical Hospital; Gernot Klein, MD, Principal Investigator — APEX GmbH; Mircea N Penescu, MD, Principal Investigator — Carol Davila Nephrology Hospital Bucharest
Locations (3):
- APEX GmbH, Munich, Germany
- Republican Clinical Hospital, Chisinau, Moldova
- Carol Davila Nephrology Hospital Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided